CLINICAL TRIAL: NCT05444504
Title: Effectiveness and Acceptability of Two Insertable Device Models for Non-surgical Management of Obstetric Fistula: a Randomized Crossover Trial
Brief Title: Effectiveness and Acceptability of Insertable Devices for Obstetric Fistula Management
Acronym: COPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Korle-Bu Teaching Hospital, Accra, Ghana (Other); Restore Health (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Gynocare Women's and Fistula Hospital, Eldorat, Kenya (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: P0555006; R01HD108236 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obstetric Fistula; Fistula; Fistula, Urinary; Fistula, Vaginal
Keywords: Menstrual cup; Urinary incontinence; Fistula; Obstetric Fistula; Fistula, Vaginal; Fistula, Urinary; Women's health; Quality of LIfe
MeSH Terms: conditions — Fistula; Urinary Fistula; Vaginal Fistula; Urinary Incontinence | interventions — Menstrual Hygiene Products

STUDY DESIGN:
Intervention Model Description: The investigators will compare two intervention models among women awaiting fistula surgery or whose surgery was unsuccessful: 1) a vaginal cup ('cup'), and 2) the cup attached via rubber tubing to a leg-secured urine collection bag ('cup+') for greater urine holding capacity (Table 1). Using a crossover design for efficiency, the investigators will randomize 100 participants to one of two sequences of leaking freely, cup, and cup+ at fistula centers in Ghana, Kenya, and Uganda, then re-randomize to continue using the cup or cup+ at home for up to 3 months. This design includes repeated measures of leakage (4 per participant, total obs=400), uses participants as their own controls, reduces the risk of confounding due to intervention order, and captures usual leaking variability through multiple measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Other): 24 hours of use each of leaking freely, leaking freely, cup, and then cup+
  Interventions: Device: Cup; Device: Cup+
- Group 2 (Other): 24 hours of use each of leaking freely, cup, cup+, and then cup
  Interventions: Device: Cup; Device: Cup+

INTERVENTIONS:
Device: Cup — an insertable vaginal cup ('cup')
Device: Cup+ — the cup attached via rubber tubing to a leg-secured urine collection bag ('cup+') for greater urine holding capacity

SUMMARY:
The investigators propose a clinical trial and nested qualitative study to 1) quantify the effectiveness of an insertable vaginal cup to manage fistula urinary incontinence, 2) examine user and implementer acceptability, and 3) quantify fistula management cost. Two intervention models will be compared among women awaiting fistula surgery or whose surgery was unsuccessful: 1) a vaginal cup ('cup'), and 2) the cup attached via rubber tubing to a leg-secured urine collection bag ('cup+') for greater urine holding capacity.

DETAILED DESCRIPTION:
Obstetric fistula is a traumatic maternal morbidity resulting in severe urinary incontinence that increases stigma and reduces quality of life. The estimated two million women with fistula, most in sub-Saharan Africa, face substantial multi-level barriers to surgical repair. Women need an acceptable non-surgical option for therapeutic management of fistula-related urinary incontinence, yet no non-surgical standard of care exists. Use of an insertable silicone vaginal cup has great potential for fistula management; it is effective for menstrual management and efficacious at reducing short-term fistula urinary leakage.

The investigators propose a clinical trial and nested qualitative study to 1) quantify the effectiveness of an insertable vaginal cup to manage fistula urinary incontinence, 2) examine user and implementer acceptability, and 3) quantify fistula management cost. Two intervention models will be compared among women awaiting fistula surgery or whose surgery was unsuccessful: 1) a vaginal cup ('cup'), and 2) the cup attached via rubber tubing to a leg-secured urine collection bag ('cup+') for greater urine holding capacity. Using a cross-over design for efficiency, 100 participants will be randomized to one of two sequences of leaking freely, cup, and cup+ at fistula centers in Ghana, Kenya, and Uganda and observed for four days (total observations=400). Each treatment (cup, cup+ or leaking freely) is used for 24h for day and night use, then crossover. Data are captured through self-report and clinical checklist. On day 4, participants are re-randomized to use cup or cup+ at home for 3 months. Acceptability assessment is informed by implementation and health behavior theory.

Aim 1. To quantify the effectiveness and comparative effectiveness of the cup and cup+. The trial will compare objective and patient-reported measures of effectiveness of the cup and cup+ to leaking freely and of the cup to the cup+. Short-term assessment will be objective (urinary leakage; 8, 24hrs), long-term assessment will be patient-reported (QoL; 1-3 months).

Aim 2. To examine acceptability of cup and cup+. User and implementer acceptability will be assessed using a sequential explanatory mixed-methods design. Acceptability among trial participants will be measured longitudinally (1-3 months). User and implementer acceptability will be examined within in-depth interviews of selected trial participants (n~30) at 3 months and potential implementers (ob/gyns, midwives/nurses, community health workers, n~20).

Aim 3. To explore the material and opportunity costs to non-surgical fistula management. Surveys and time motion study among trial participants at facility and community will estimate direct and indirect costs of fistula management from a patient perspective. The long-term goal of the proposed work is to overcome barriers to comprehensive fistula care and increase quality of life through an acceptable, non-surgical option for therapeutic management of fistula.

ELIGIBILITY:
Inclusion criteria:

* VVF confirmed by dye test and clinical exam at least 3cm from the external urethral orifice (regardless of size), adequate vaginal capacity to accommodate the cup (per physician)
* Willing to insert and remove cup/cup+
* Clear understanding of the study procedures
* Willing to participate fully, not yet been repaired or previously failed surgical repair, at least 6mo post-surgery
* If previous fistula repair, ≥3mo post-delivery
* If recent birth, age 18+ or emancipated minor
* Speak English or local language

Exclusion criteria:

* Any rectovaginal fistula
* Urinary leakage <6ml over 6 hours
* Women who are candidates for catheterization who could be healed without surgery will be excluded as they are <3mo post-delivery.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in volume of observed urine leakage | baseline to 6 hours
  Urine leakage will be measured in mL using pad weight

SECONDARY OUTCOMES:
Mean change in volume of perceived urine leakage | baseline vs. 6 hours, 24 hours,1 month, 2 months and 3 months
  Perceived urine leakage will be measured by the International Consultation on Incontinence Questionnaire SF (ICIQ-SF). This score ranges from 0-21 with higher scores indicating greater incontinence.
Mean change in WHO Quality of Life BREF (WHOQOL-BREF) score | baseline vs. 24 hours, 1 month, 2 months and 3 months
  Quality of life will be measured using the WHOQOL-BREF. The score ranges from 0-100 with higher scores indicating higher quality of life.
Mean change in fistula-related stigma scale | baseline vs. 1 month, 2 months and 3 months
  Stigma will be measured using the fistula-related stigma scale, and enacted and internalized subscales. This score ranges from 0-100 with higher scores indicating higher stigma.
Mean change in fistula management costs over time | baseline vs. 1 month, 2 months, and 3 months
  Fistula management costs will be calculated by combining the total material costs and lost wages in Ghanaian Cedi (local currency) over time. Time in minutes will inform calculations of lost wages using prevailing wage rates for the study population. The mean change in cost will be from baseline to 3 months.
Mean change in sleep satisfaction using the WHO sleep index | baseline vs. 1 month, 2 months, and 3 months
  Sleep satisfaction using the adapted WHO sleep index. The score ranges from 1-5 where 1 is least satisfied and 5 is very satisfied.
Mean change in Coping Orientation to Problems Experienced Inventory (BRIEF) Coping scale | baseline vs. 1 month, 2 months, and 3 months
  Coping will be measured using the modified BRIEF Coping scale. The score ranges from 0-100 with higher scores indicating better coping.
Mean change in perceived empowerment over time | baseline vs. 1 month, 2 months, and 3 months
  Empowerment change in the proportion of users across physical mobility, participation in income-generating activities, bodily autonomy, household decision making, reproductive autonomy, and social participation. Individual measures will be captured using a scale of 1-5, with 1 indicating lower empowerment and 5 higher.
Changes in perceived safety over time | baseline vs. 6 hours, 24 hours, 1 month, 2 months, and 3 months
  change in the proportion of users who report any adverse events with use of the intervention model at 1, 2, and 3-month follow up
Changes in user acceptability of the intervention over time | 6 hours vs. 24 hours, 1 month, 2 months, and 3 months
  Proportion of users who report the intervention as acceptable measured across domains including easy to insert, remove, clean, comfortable to wear, interference with activities, perceived efficacy, self-efficacy, intent to use, and reported using a mean acceptability scale (based on composite score of acceptability items) regarding the intervention model. Standardized range will be 0-100, with higher values meaning greater acceptability and lower values lower acceptability.
Changes in post-fistula repair reintegration scale | baseline vs. 1 month, 2 months, and 3 months
  Reintegration will be measured using the post-fistula repair reintegration scale and subdomains comfort with relatives, relationship, general life satisfaction, family needs, and social engagement. The score ranges from 0-100 with higher scores indicating higher reintegration/functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Alison El Ayadi, ScD, Principal Investigator — University of California, San Francisco; Nessa Ryan, PhD, Study Director — Restore Health
Locations (3):
- Ghana (2):
  - Mercy Women's Catholic Hospital, Mankessim
  - Tamale Fistula Center, Tamale
- Gynocare Women's and fistula hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data will be deidentified and made available after all study publications have been completed without cost to researchers and analysts. Qualitative data and associated documentation will be available to users under a data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after primary and secondary analyses have been completed.
Access Criteria: Data access requests should include 1) Indicate title of their study, a brief rationale for the proposal, the methods of analysis, and the inclusion and exclusion criteria; 2) Include the approval of their Institutional Review Board/ Committee on Human Research; 3) Indicate what they plan to do with the data; 4) Include assurances that they will not share the data with others without the written permission of Dr. El Ayadi; 5) Commit to using the data only for research purposes; 6) Commit to securing the data using appropriate computer technology; 7) Commit to destroying or returning the data after analyses are completed, and; 8) Agree to give proper credit in any publications resulting from the data via citation of the grant and the investigators who obtained the data. Researchers will have to sign a Data Use Agreement that includes these terms, as well as a commitment that they will not attempt to identify individual respondents.
URL: http://datadryad.org

REFERENCES:
- [Background] Wall LL. Obstetric vesicovaginal fistula as an international public-health problem. Lancet. 2006 Sep 30;368(9542):1201-9. doi: 10.1016/S0140-6736(06)69476-2. PMID 17011947
- [Background] De Ridder D. Vesicovaginal fistula: a major healthcare problem. Curr Opin Urol. 2009 Jul;19(4):358-61. doi: 10.1097/MOU.0b013e32832ae1b7. PMID 19440154
- [Background] Adler AJ, Ronsmans C, Calvert C, Filippi V. Estimating the prevalence of obstetric fistula: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2013 Dec 30;13:246. doi: 10.1186/1471-2393-13-246. PMID 24373152
- [Background] Tebeu PM, Fomulu JN, Khaddaj S, de Bernis L, Delvaux T, Rochat CH. Risk factors for obstetric fistula: a clinical review. Int Urogynecol J. 2012 Apr;23(4):387-94. doi: 10.1007/s00192-011-1622-x. Epub 2011 Dec 6. PMID 22143450
- [Background] GHS. Report on Fistula Burden in Ghana. 2015.
- [Background] Barageine JK, Beyeza-Kashesya J, Byamugisha JK, Tumwesigye NM, Almroth L, Faxelid E. "I am alone and isolated": a qualitative study of experiences of women living with genital fistula in Uganda. BMC Womens Health. 2015 Sep 10;15:73. doi: 10.1186/s12905-015-0232-z. PMID 26359255
- [Background] Mwini-Nyaledzigbor PP, Agana AA, Pilkington FB. Lived experiences of Ghanaian women with obstetric fistula. Health Care Women Int. 2013;34(6):440-60. doi: 10.1080/07399332.2012.755981. PMID 23641897
- [Background] Tellier S, Hyttel M. Menstrual Health Management in East and Southern Africa: a Review Paper. United Nations Population Fund and WoMena; 2018.
- [Background] Baker Z, Bellows B, Bach R, Warren C. Barriers to obstetric fistula treatment in low-income countries: a systematic review. Trop Med Int Health. 2017 Aug;22(8):938-959. doi: 10.1111/tmi.12893. Epub 2017 Jul 20. PMID 28510988
- [Background] Banke-Thomas AO, Wilton-Waddell OE, Kouraogo SF, Mueller E. Current evidence supporting obstetric fistula prevention strategies in sub Saharan Africa: a systematic review of the literature. Afr J Reprod Health. 2014 Sep;18(3):118-27. PMID 25438516
- [Background] Fernandez-Romero JA, Deal C, Herold BC, Schiller J, Patton D, Zydowsky T, Romano J, Petro CD, Narasimhan M. Multipurpose prevention technologies: the future of HIV and STI protection. Trends Microbiol. 2015 Jul;23(7):429-436. doi: 10.1016/j.tim.2015.02.006. Epub 2015 Mar 7. PMID 25759332
- [Background] North BB, Oldham MJ. Preclinical, clinical, and over-the-counter postmarketing experience with a new vaginal cup: menstrual collection. J Womens Health (Larchmt). 2011 Feb;20(2):303-11. doi: 10.1089/jwh.2009.1929. Epub 2011 Jan 1. PMID 21194348
- [Background] Beksinska ME, Smit J, Greener R, Todd CS, Lee ML, Maphumulo V, Hoffmann V. Acceptability and performance of the menstrual cup in South Africa: a randomized crossover trial comparing the menstrual cup to tampons or sanitary pads. J Womens Health (Larchmt). 2015 Feb;24(2):151-8. doi: 10.1089/jwh.2014.5021. PMID 25682816
- [Background] Hyttel M, Thomsen CF, Luff B, Tellier M, Storrusten H, Nyakato VN. Drivers and challenges to use of menstrual cups among schoolgirls in rural Uganda: A qualitative study. Waterlines. 2017;36(2):109-24.
- [Background] Russell KW, Robinson RE, Mone MC, Scaife CL. Enterovaginal or Vesicovaginal Fistula Control Using a Silicone Cup. Obstet Gynecol. 2016 Dec;128(6):1365-1368. doi: 10.1097/AOG.0000000000001745. PMID 27824744
- [Background] Goldberg L, Elsamra S, Hutchinson-Colas J, Segal S. Delayed Diagnosis of Vesicouterine Fistula After Treatment for Mixed Urinary Incontinence: Menstrual Cup Management and Diagnosis. Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):e29-31. doi: 10.1097/SPV.0000000000000301. PMID 27403759
- [Background] New Vision Reporter. Menstrual cup: Temporary relief for fistula patients. New Vision. 2012.
- [Background] Ganyaglo GYK, Ryan N, Park J, Lassey AT. Feasibility and acceptability of the menstrual cup for non-surgical management of vesicovaginal fistula among women at a health facility in Ghana. PLoS One. 2018 Nov 28;13(11):e0207925. doi: 10.1371/journal.pone.0207925. eCollection 2018. PMID 30485344
- [Background] Shaw C, Logan K, Webber I, Broome L, Samuel S. Effect of clean intermittent self-catheterization on quality of life: a qualitative study. J Adv Nurs. 2008 Mar;61(6):641-50. doi: 10.1111/j.1365-2648.2007.04556.x. PMID 18302605
- [Background] Wilde MH, Fader M, Ostaszkiewicz J, Prieto J, Moore K. Urinary bag decontamination for long-term use: a systematic review. J Wound Ostomy Continence Nurs. 2013 May-Jun;40(3):299-308. doi: 10.1097/WON.0b013e3182800305. PMID 23652701
- [Background] Wilde MH. Life with an indwelling urinary catheter: the dialectic of stigma and acceptance. Qual Health Res. 2003 Nov;13(9):1189-204. doi: 10.1177/1049732303257115. PMID 14606409
- [Background] Avery M, Prieto J, Okamoto I, Cullen S, Clancy B, Moore KN, Macaulay M, Fader M. Reuse of intermittent catheters: a qualitative study of IC users' perspectives. BMJ Open. 2018 Aug 17;8(8):e021554. doi: 10.1136/bmjopen-2018-021554. PMID 30121601
- [Background] Prieto J, Murphy CL, Moore KN, Fader M. Intermittent catheterisation for long-term bladder management. Cochrane Database Syst Rev. 2014 Sep 10;(9):CD006008. doi: 10.1002/14651858.CD006008.pub3. PMID 25208303
- [Background] Wyndaele JJ, Brauner A, Geerlings SE, Bela K, Peter T, Bjerklund-Johanson TE. Clean intermittent catheterization and urinary tract infection: review and guide for future research. BJU Int. 2012 Dec;110(11 Pt C):E910-7. doi: 10.1111/j.1464-410X.2012.11549.x. Epub 2012 Oct 4. PMID 23035877
- [Background] Madersbacher H. The Dilemma With the Terminology and the Studies of Intermittent Catheterization: What Is the Best Course of Action? Current Bladder Dysfunction Reports. 2017;12(4):349-53.
- [Background] Chapple A, Prinjha S, Feneley R, Ziebland S. Drawing on Accounts of Long-Term Urinary Catheter Use: Design for the "Seemingly Mundane". Qual Health Res. 2016 Jan;26(2):154-63. doi: 10.1177/1049732315570135. Epub 2015 Feb 2. PMID 25646001
- [Background] Okoye UO, Emma-Echiegu N, Tanyi PL. Living with vesico-vaginal fistula: experiences of women awaiting repairs in Ebonyi State, Nigeria. Tanzan J Health Res. 2014 Oct;16(4):322-8. doi: 10.4314/thrb.v16i4.9. PMID 26891522
- [Background] Ryan N. Stigma and coping among women living with obstetric fistula in Ghana: a mixed methods study. New York: New York University College of Global Public Health; 2019.
- [Background] Mantey R, Kotoh AM, Barry M, Redington W. Womens' experiences of living with obstetric fistula in Ghana-time for the establishment of a fistula centre of excellence. Midwifery. 2020 Mar;82:102594. doi: 10.1016/j.midw.2019.102594. Epub 2019 Dec 13. PMID 31874317
- [Background] Changole J, Thorsen VC, Kafulafula U. "I am a person but I am not a person": experiences of women living with obstetric fistula in the central region of Malawi. BMC Pregnancy Childbirth. 2017 Dec 21;17(1):433. doi: 10.1186/s12884-017-1604-1. PMID 29268711
- [Background] Epiu I, Alia G, Mukisa J, Tavrow P, Lamorde M, Kuznik A. Estimating the cost and cost-effectiveness for obstetric fistula repair in hospitals in Uganda: a low income country. Health Policy Plan. 2018 Nov 1;33(9):999-1008. doi: 10.1093/heapol/czy078. PMID 30252051
- [Background] Keya KT, Sripad P, Nwala E, Warren CE. "Poverty is the big thing": exploring financial, transportation, and opportunity costs associated with fistula management and repair in Nigeria and Uganda. Int J Equity Health. 2018 Jun 1;17(1):70. doi: 10.1186/s12939-018-0777-1. PMID 29859118
- [Background] Brook G, Tessema AB. Obstetric fistula: the use of urethral plugs for the management of persistent urinary incontinence following successful repair. Int Urogynecol J. 2013 Mar;24(3):479-84. doi: 10.1007/s00192-012-1887-8. Epub 2012 Jul 18. PMID 22806488
- [Background] Norton JM, Dodson JL, Newman DK, Rogers RG, Fairman AD, Coons HL, Star RA, Bavendam TG. Nonbiologic factors that impact management in women with urinary incontinence: review of the literature and findings from a National Institute of Diabetes and Digestive and Kidney Diseases workshop. Int Urogynecol J. 2017 Sep;28(9):1295-1307. doi: 10.1007/s00192-017-3400-x. Epub 2017 Jul 3. PMID 28674734
- [Background] Debas HT, Donkor P, Gawande A, Jamison DT, Kruk ME, Mock CN, editors. Essential Surgery: Disease Control Priorities, Third Edition (Volume 1). Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2015 Apr 2. Available from http://www.ncbi.nlm.nih.gov/books/NBK333500/ PMID 26740991
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Creswell J, Plano Clark V. Designing and Conducting Mixed Methods Research. 2nd ed: Sage Publications, Inc; 2011.
- [Background] Wellek S, Blettner M. On the proper use of the crossover design in clinical trials: part 18 of a series on evaluation of scientific publications. Dtsch Arztebl Int. 2012 Apr;109(15):276-81. doi: 10.3238/arztebl.2012.0276. Epub 2012 Apr 13. PMID 22567063
- [Background] El Ayadi AM, Barageine J, Korn A, Kakaire O, Turan J, Obore S, Byamugisha J, Lester F, Nalubwama H, Mwanje H, Tripathi V, Miller S. Trajectories of women's physical and psychosocial health following obstetric fistula repair in Uganda: a longitudinal study. Trop Med Int Health. 2019 Jan;24(1):53-64. doi: 10.1111/tmi.13178. Epub 2018 Nov 18. PMID 30372572
- [Background] Webster J, Nicholas C, Velacott C, Cridland N, Fawcett L. Validation of the WHOQOL-BREF among women following childbirth. Aust N Z J Obstet Gynaecol. 2010 Apr;50(2):132-7. doi: 10.1111/j.1479-828X.2009.01131.x. PMID 20522068
- [Background] Juma J, Nyothach E, Laserson KF, Oduor C, Arita L, Ouma C, Oruko K, Omoto J, Mason L, Alexander KT, Fields B, Onyango C, Phillips-Howard PA. Examining the safety of menstrual cups among rural primary school girls in western Kenya: observational studies nested in a randomised controlled feasibility study. BMJ Open. 2017 May 4;7(4):e015429. doi: 10.1136/bmjopen-2016-015429. PMID 28473520
- [Background] NCAA. A Factsheet for Student Athletes: Assess Your Hydration Status. 2017.
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Gale NK, Heath G, Cameron E, Rashid S, Redwood S. Using the framework method for the analysis of qualitative data in multi-disciplinary health research. BMC Med Res Methodol. 2013 Sep 18;13:117. doi: 10.1186/1471-2288-13-117. PMID 24047204
- [Background] van Eijk AM, Zulaika G, Lenchner M, Mason L, Sivakami M, Nyothach E, Unger H, Laserson K, Phillips-Howard PA. Menstrual cup use, leakage, acceptability, safety, and availability: a systematic review and meta-analysis. Lancet Public Health. 2019 Aug;4(8):e376-e393. doi: 10.1016/S2468-2667(19)30111-2. Epub 2019 Jul 16. PMID 31324419
- [Background] Pope R. Research in Obstetric Fistula: Addressing Gaps and Unmet Needs. Obstet Gynecol. 2018 May;131(5):863-870. doi: 10.1097/AOG.0000000000002578. PMID 29630017
- [Background] U.S. Department of Health and Human Services NIoH, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1. July 2017 [Available from: https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf.
- [Background] Imoto A, Matsuyama A, Ambauen-Berger B, Honda S. Health-related quality of life among women in rural Bangladesh after surgical repair of obstetric fistula. Int J Gynaecol Obstet. 2015 Jul;130(1):79-83. doi: 10.1016/j.ijgo.2015.01.018. Epub 2015 Apr 20. PMID 25935472
- [Background] El Ayadi A, Nalubwama H, Barageine J, Neilands TB, Obore S, Byamugisha J, Kakaire O, Mwanje H, Korn A, Lester F, Miller S. Development and preliminary validation of a post-fistula repair reintegration instrument among Ugandan women. Reprod Health. 2017 Sep 2;14(1):109. doi: 10.1186/s12978-017-0372-8. PMID 28865473
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Derived] Ryan N, Ganyaglo GYK, Park J, Lin TK, Pozen J, Mittal A, El Ayadi AM. Effectiveness and acceptability of two insertable device models for non-surgical management of obstetric fistula: protocol for a hybrid type I randomized crossover trial. BMC Womens Health. 2025 Jul 4;25(1):314. doi: 10.1186/s12905-025-03823-y. PMID 40615875